CLINICAL TRIAL: NCT06126224
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of KarXT for the Treatment of Psychosis Associated With Alzheimer's Disease
Brief Title: A Study to Assess Efficacy and Safety of KarXT for the Treatment of Psychosis Associated With Alzheimer's Disease (ADEPT-2)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN012-0027; KAR-032 (Other: Karuna Pharmaceuticals Protocol ID); CN012-0027 (Other: Bristol-Myers Squibb Protocol ID)
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Psychosis Associated With Alzheimer's Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT (Experimental): Xanomeline and Trospium Chloride Capsules
  Interventions: Drug: KarXT
- Placebo (Placebo Comparator): Placebo Capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KarXT — KarXT 20/2 mg (total daily dose [TDD] 60/6 mg) KarXT 30/3 mg (TDD 90/9 mg) KarXT 40/4 mg (TDD 120/12 mg) KarXT 50/5 mg (TDD 150/15 mg) KarXT 66.7/6.67 mg (TDD 200/20 mg)
  Arms: KarXT
Drug: Placebo — Placebo Capsules
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, double-blind, placebo-controlled, parallel group study to evaluate the safety and efficacy of KarXT in male and female subjects who are aged 55 to 90 years and have mild to severe Alzheimer's Disease (AD) with moderate to severe psychosis related to AD.

The primary objective of the study is to evaluate the efficacy of KarXT compared with placebo in the treatment of subjects with psychosis associated with AD as measured by the Neuropsychiatric Inventory-Clinician (NPI-C): Hallucinations and Delusions (H+D) score.

ELIGIBILITY:
Key Inclusion Criteria:

1. Is a male or female aged 55 to 90 years, inclusive, at Screening.
2. Can understand the nature of the trial and protocol requirements and provide informed consent or assent before any study assessments are performed.
3. Meets clinical criteria for Possible AD or Probable AD.
4. Living at the same home or residential assisted-living facility for a minimum of 6 weeks before Screening.
5. Have an identified study partner who should have daily contact (approximately 10 hours a week or more).
6. History of psychotic symptoms (meeting International Psychogeriatric Association criteria) (Cummings 2020) for at least 2 months prior to Screening.
7. CGI-S scale with a score ≥ 4 at Screening and Baseline.
8. AD subjects are required to have NPI-C: Hallucinations and Delusions (H+D) score of ≥ 6 AND meet at least 1 of the following criteria at Screening and Baseline:

   1. Moderate to severe delusions, defined as NPI-C: Delusions domain score of ≥ 2 on 2 of the 8 items OR
   2. Moderate to severe hallucinations, defined as NPI-C: Hallucinations domain score of ≥ 2 on 2 of the 7 items
9. MMSE score of 8 to 22, inclusive, at Screening.

Key Exclusion Criteria:

1. Psychotic symptoms that are primarily attributable to a condition other than the AD causing the dementia.
2. History of major depressive episode with psychotic features during the 12 months prior to Screening.
3. History of bipolar disorder, schizophrenia, or schizoaffective disorder.
4. Significant or severe medical conditions including pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, cardiovascular, or oncologic disease or any other condition that, in the opinion of the Investigator, could jeopardize the safety of the subject, ability to complete or comply with the study procedures or validity of the study results.
5. History or high risk of urinary retention, gastric retention, or narrow-angle glaucoma as evaluated by the Investigator.
6. Prior exposure to KarXT.
7. History of hypersensitivity to KarXT excipients or trospium chloride.
8. Experienced any significant adverse events (AEs) due to trospium.
9. Participation in another clinical study in which the subject received an experimental or investigational drug within 3 months before Screening or has participated in more than 2 clinical studies in the 12 months prior to Screening.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to End of Treatment in the Neuropsychiatric Inventory-Clinician: Hallucinations and Delusions (NPI-C: H+D) score | Baseline and End of Treatment (up to 14 weeks)
  Neuropsychiatric Inventory-Clinician: Hallucinations and Delusions scale includes 2 domains from the NPI-C scale, namely, hallucinations and delusions. These 2 domains include the following number of items to be rated by the clinician: Hallucinations, 7 items (maximum score = 21) and Delusions, 8 items (maximum score = 24). The maximum score for the NPI-C: H+D scale is 45. Higher scores on this scale indicate worse outcomes.

SECONDARY OUTCOMES:
Change from Baseline to End of Treatment in the Cohen-Mansfield Agitation Inventory (CMAI) score | Baseline and End of Treatment (up to 14 weeks)
  Cohen-Mansfield Agitation Inventory (CMAI) is a caregiver's rating 29-item questionnaire used to assess the frequency of manifestations of agitated behaviors in older adults. Each item is rated on a 7-point scale ranging from "1 = never" to "7 = several times per hour." Higher scores on this scale indicate worse outcomes.
Change from Baseline to End of Treatment in the Clinical Global Impressions-Severity (CGI-S) scale | Baseline and End of Treatment (up to 14 weeks)
  Clinical Global Impressions-Severity (CGI-S) requires the assessor to consider aspects of the psychosis (hallucinations and delusions) prior to providing a global assessment of severity. Higher scores on this scale indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (119):
- United States (61):
  - Local Institution - 1116, Chandler, Arizona
  - Local Institution - 1044, Phoenix, Arizona
  - Local Institution - 1104, Anaheim, California
  - Local Institution - 1119, Canoga Park, California
  - Local Institution - 1151, Encino, California
  - Local Institution - 1142, Lancaster, California
  - Local Institution - 1117, Los Alamitos, California
  - Local Institution - 1103, Sherman Oaks, California
  - Local Institution - 1007, Walnut Creek, California
  - Local Institution - 1156, Clermont, Florida
  - Local Institution - 1138, Cutler Bay, Florida
  - Local Institution - 1162, Delray Beach, Florida
  - Local Institution - 1164, Doral, Florida
  - Local Institution - 1165, Fort Myers, Florida
  - Local Institution - 1155, Hialeah, Florida
  - Local Institution - 1107, Hialeah, Florida
  - Local Institution - 1120, Hialeah, Florida
  - Local Institution - 1140, Hialeah, Florida
  - Local Institution - 0150, Homestead, Florida
  - Local Institution - 1145, Homestead, Florida
  - Local Institution - 1127, Largo, Florida
  - Local Institution - 1039, Maitland, Florida
  - Local Institution - 1146, Maitland, Florida
  - Local Institution - 1159, Miami, Florida
  - Local Institution - 1118, Miami, Florida
  - Local Institution - 1111, Miami, Florida
  - Local Institution - 1108, Miami, Florida
  - Local Institution - 1125, Miami, Florida
  - Local Institution - 1115, Miami, Florida
  - Local Institution - 1143, Miami, Florida
  - Local Institution - 1113, Miami, Florida
  - Local Institution - 1009, Miami, Florida
  - Local Institution - 1129, Miami, Florida
  - Local Institution - 1150, Miami, Florida
  - Local Institution - 1109, Miami, Florida
  - Local Institution - 1158, Miami, Florida
  - Local Institution - 1147, Miami, Florida
  - Local Institution - 1105, Miami, Florida
  - Local Institution - 1157, Miami, Florida
  - Local Institution - 1126, Miami Gardens, Florida
  - Local Institution - 1102, Miami Lakes, Florida
  - Local Institution - 1101, Okeechobee, Florida
  - Local Institution - 1136, Orlando, Florida
  - Local Institution - 1112, Orlando, Florida
  - Local Institution - 1137, Port Orange, Florida
  - Local Institution - 1133, Sweetwater, Florida
  - Local Institution - 1041, Tampa, Florida
  - Local Institution - 1124, Tampa, Florida
  - Local Institution - 1123, Tampa, Florida
  - Local Institution - 1110, Tampa, Florida
  - Local Institution - 1131, Viera, Florida
  - Local Institution - 1161, Decatur, Georgia
  - Local Institution - 1148, Elgin, Illinois
  - Local Institution - 1114, Marrero, Louisiana
  - Local Institution - 1139, Rochester Hills, Michigan
  - Local Institution - 1132, Flowood, Mississippi
  - Local Institution - 1122, Dayton, Ohio
  - Local Institution - 1106, Cypress, Texas
  - Local Institution - 1163, Houston, Texas
  - Local Institution - 1154, Katy, Texas
  - Local Institution - 1134, Stafford, Texas
- Belgium (3):
  - Local Institution - 2801, Hasselt, Limburg
  - Local Institution - 2802, Leuven, Vlaams Brabant
  - Local Institution - 2803, Roeselare, West-Vlaanderen
- Chile (3):
  - Local Institution - 6002, Providencia, Santiago Metropolitan
  - Local Institution - 6003, Antofagasta
  - Local Institution - 6001, Las Condes
- China (19):
  - Local Institution - 7007, Hefei, Anhui
  - Local Institution - 7004, Beijing, Beijing Municipality
  - Local Institution - 7005, Beijing, Beijing Municipality
  - Local Institution - 7015, Chongqing, Chongqing Municipality
  - Local Institution - 7008, Guangzhou, Guangdong
  - Local Institution - 7016, Guangzhou, Guangdong
  - Local Institution - 7009, Guangzhou, Guangdong
  - Local Institution - 7003, Shenzhen, Guangdong
  - Local Institution - 7013, Nanjing, Jiangsu
  - Local Institution - 7012, Nanchang, Jiangxi
  - Local Institution - 7001, Shanghai, Shanghai Municipality
  - Local Institution - 7011, Shanghai, Shanghai Municipality
  - Local Institution - 7002, Chengdu, Sichuan
  - Local Institution - 7019, Tianjin, Tianjin Municipality
  - Local Institution - 7017, Hangzhou, Zhejiang
  - Local Institution - 7010, Hangzhou, Zhejiang
  - Local Institution - 7006, Hangzhou, Zhejiang
  - Local Institution - 7020, Hangzhou, Zhejiang
  - Local Institution - 7018, Wenzhou, Zhejiang
- Greece (5):
  - Local Institution - 4805, Athens, Attica
  - Local Institution - 4803, Athens, Attica
  - Local Institution - 4802, Chaidari, Athens, Attica
  - Local Institution - 4806, Marousi, Attica
  - Local Institution - 4801, Heraklion
- Hungary (3):
  - Local Institution - 4601, Pécs, Baranya
  - Local Institution - 4602, Budapest
  - Local Institution - 4603, Miskolc
- Mexico (5):
  - Local Institution - 1502, Saltillo Centro, Coahuila
  - Local Institution - 1503, Monterrey, Nuevo León
  - Local Institution - 1505, Monterrey, Nuevo León
  - Local Institution - 1501, Culiacán, Sinaloa
  - Local Institution - 1506, México
- Local Institution - 6103, Pueblo Libre, Lima region, Peru
- Poland (7):
  - Local Institution - 4206, Lublin, Lublin Voivodeship
  - Local Institution - 4207, Lodz, Lódzkie
  - Local Institution - 4208, Katowice, Silesian Voivodeship
  - Local Institution - 4204, Bydgoszcz
  - Local Institution - 4205, Katowice
  - Local Institution - 4202, Lodz
  - Local Institution - 4201, Ścinawa
- South Korea (7):
  - Local Institution - 7208, Buk-gu, Daegu Gwang'yeogsi
  - Local Institution - 7207, Seongnam-si, Gyeonggido
  - Local Institution - 7205, Incheon, Incheon Gwang'yeogsi
  - Local Institution - 7202, Seongnam-si
  - Local Institution - 7206, Seoul
  - Local Institution - 7203, Seoul
  - Local Institution - 7201, Seoul
- Turkey (Türkiye) (5):
  - Local Institution - 4702, Atakum, Samsun
  - Local Institution - 4701, Eskişehir
  - Local Institution - 4704, Istanbul
  - Local Institution - 4705, Izmir
  - Local Institution - 4703, Izmir

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06126224.html